CLINICAL TRIAL: NCT00478881
Title: Randomized, Double-blind, Placebo-controlled, Parallel Group Study of Vardenafil 10 mg Twice Daily to Assess the Effect on Urodynamics in Patients With Overactive Bladder (Detrusor Overactivity)
Brief Title: A Study To Assess If 10 mg Vardenafil (BAY38-9456) Taken Twice Daily For 6 Weeks Has An Effect On Bladder Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12392; 2006-005145-11 (EudraCT Number)
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Results first posted 2009-12-24 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-11

CONDITIONS: Overactive Bladder; Detrusor Overactivity
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vardenafil HCl (Levitra, BAY38-9456) (Experimental): vardenafil hydrochloride 10 mg film-coated tablets twice daily (BID) for oral (by mouth) intake for 6 weeks
  Interventions: Drug: Vardenafil HCl (Levitra, BAY38-9456)
- Placebo (Placebo Comparator): vardenafil hydrochloride-matching film-coated tablets BID for oral intake for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil HCl (Levitra, BAY38-9456) — vardenafil hydrochloride 10 mg film-coated tablets twice daily (BID) for oral (by mouth) intake for 6 weeks
  Arms: Vardenafil HCl (Levitra, BAY38-9456)
Drug: Placebo — vardenafil hydrochloride-matching film-coated tablets BID for oral intake for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess if the study drug, Vardenafil (approved by Health Authorities is available on the market for treatment of erectile dysfunction) has an effect on bladder function and micturition frequency. The study drug is to be taken in the form of tablets twice a day, one tablet in the morning and one tablet in the evening. A non-active treatment (placebo), a sugar pill, will be used as a comparator to see if the new study drug works better than no drug. The timing of visits for the study is as follows: the 1st visit (screening visit) at beginning of run-in-assessment with qualifying tests for patients: electrocardiogram (ECG), safety laboratory and residual urine (by ultrasonography: a non-invasive examination using ultrasound for the assessment of the bladder). 2nd visit (randomization visit). During visit this should be performed: urodynamic measurements (filling cystometry and pressure flow investigations), ECG and safety laboratory. 3rd visit (safety visit) takes place at two up to three weeks of randomized treatment. 4th visit (final visit)-following test should be done: urodynamic measurements (filling cystometry and pressure flow investigations), ECG, safety laboratory and residual urine (by ultrasonography); A phone call 24 hours after visit 4 to assess any SAEs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged > 18 years (females either postmenopausal or using adequate birth control)
* Urodynamic criteria:

  * Entire bladder capacity (= maximum cystometric bladder capacity) < 300 mL OR
  * In accordance with International Continence Society (ICS)-guidelines: Detrusor overactivity as defined as spontaneous involuntary detrusor contraction during filling phase OR
  * Detrusor contraction during filling phase leading to involuntarily initiated micturition before a normal bladder capacity is reached
* Patient micturition diary criteria: at least 8 micturitions per day AND at least 1 urgency episode per day
* Signed and dated written Patient Informed Consent Form

Exclusion Criteria:

* Treatment with drugs known to affect urinary bladder function
* Known other reasons for micturition problems than detrusor overactivity
* Recent intervention in urogenital tract
* Abnormal liver or renal lab values
* Treatment with nitrates or nitric oxide donors, alpha-blockers, potent inhibitors of CYP-450 3A4, acenocoumarol, heparin, drugs known to prolong QT-interval
* NAION, hereditary regenerative retinal disorders, severe cardiovascular conditions, recent history of myocardial infarction/stroke/life-threatening arrhythmia
* congenital QT-prolongation, left ventricular outflow obstruction, severe hypo- or hypertension, symptomatic postural hypotension
* History of positive test for Hepatitis B surface antigen (HBsAg) or Hepatitis C
* Significant active peptic ulceration
* Severe chronic or acute liver disease, history of moderate (Child-Pugh B) or severe (Child-Pugh C) hepatic impairment
* In men: Clinically significant chronic haematological disease which may lead to priapism
* History of malignancy of any organ system within the past 5 years
* Bleeding disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2007-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (45):
- Bruxelles - Brussel, Belgium
- Canada (4):
  - Victoria, British Columbia
  - Brantford, Ontario
  - Kitchener, Ontario
  - Montreal, Quebec
- Czechia (2):
  - Olomouc
  - Prague
- Paris, France
- Germany (12):
  - Emmendingen, Baden-Wurttemberg
  - Bad Griesbach-Therme, Bavaria
  - Weiden, Bavaria
  - Schwedt, Brandenburg
  - Greifswald, Mecklenburg-Vorpommern
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Neunkirchen, Saarland
  - Leipzig, Saxony
  - Berlin, State of Berlin
- Budapest, Hungary
- Israel (3):
  - Haifa, Israel
  - Jerusalem, Israel
  - Petah Tikva, Israel
- Netherlands (5):
  - Eindhoven, North Brabant
  - Amsterdam
  - Maastricht
  - Rotterdam
  - Utrecht
- Poland (4):
  - Bydgoszcz
  - Chorzów
  - Siedlce
  - Warsaw
- Portugal (4):
  - Amadora
  - Lisbon
  - Porto
  - S. Martinho Do Bispo
- Russia (2):
  - Moscow
  - Saint Petersburg
- Spain (5):
  - Santiago de Compostela, A Coruña
  - Barcelona, Barcelona
  - Granada, Granada
  - Madrid, Madrid
  - Valencia, Valencia
- Basel, Canton of Basel-City, Switzerland

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started on 31 August 2007 and the last study visit occurred on 13 November 2008. The study was conducted at 56 centers in 13 countries: 45 centers in Europe, 4 centers in Canada, 4 centers in Russia, and 3 centers in Israel.
Pre-assignment Details: Number of participants screened: 635. Number of participants enrolled and randomized (started Overall study): 397. Number of participants who had taken at least one dose (Safety population): 396.
Period: Overall Study
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Started | 199 | 198
Received Medication | 198 | 198
Completed | 160 | 176
Not Completed | 39 | 22
Not completed — Adverse Event | 31 | 12
Not completed — Lack of Efficacy | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Non-Compliance with Study Medication | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo | Total
Number analyzed (Participants) | 198 | 198 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (14.2) | 58.3 (12.8) | 56.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender and age are given for those subjects who received treatment (Safety population).
  Participants
    Female | 116 | 113 | 229
    Male | 82 | 85 | 167

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bladder Volume at First Detrusor Contraction at 6 Weeks
Description: Bladder volume was measure by means of urodynamic assessments (cystometry) for up to 6 weeks. Missing data were imputed with last observation carried forward (LOCF).
Time Frame: baseline and up to 6 weeks of treatment Last Observation Carried Forward (LOCF)
Population: Modified intention-to-treat (mITT): participants included in the safety sample (received at least one dose), randomized correctly according to the Urodynamic Adjudication Board (UDAB), having one valid baseline and one valid (UDAB) on treatment urodynamic measurement. The number is not identical to participants who "completed" the study.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 122 | 136
mL | 44.993 (9.2774) | 36.948 (8.7786)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; Countries were pooled into 2 clusters, which allowed for testing of Treatment by Center interaction. An ANCOVA including Baseline (Visit 2) as a covariate with main effects for treatment and country (see pooling above) was used to test treatment difference for the primary variable and co-primary variable; Test type: Superiority or Other; p = 0.5293, ANCOVA — Bladder volume (mL) at first detrusor contraction tested first. If significant, the change in the average number of daily micturitions was to be tested using a P<0.05; Mean Difference (Final Values) = -8.045, 95% CI [-33.194 to 17.104] — Placebo-Vardenafil

2. Primary Outcome: Change From Baseline in Average Number of Daily Micturitions at 6 Weeks
Description: Change from baseline in the number of daily micturitions (bladder voidings), as reported in the participant diaries for up to 6 weeks. Missing data were imputed with last observation carried forward (LOCF).
Time Frame: baseline and up to 6 weeks of treatment LOCF
Population: Intent-to-treat (ITT) population: all randomized participants with at least one study drug medication were to be included provided they had a baseline measurement (if scheduled) and a follow-up measurement in any clinical variable. The number is not identical to participants who "completed".
Measure: Least Squares Mean (Standard Error); unit: micturitions per day
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 163 | 178
micturitions per day | -2.247 (0.2530) | -1.579 (0.2431)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0575, ANCOVA — Bladder volume (mL) at first detrusor contraction tested first. If significant, the change in the average number of daily micturitions was to be tested using a P <0.05; Mean Difference (Final Values) = 0.668, 95% CI [-0.021 to 1.358] — Placebo - Vardenafil

3. Secondary Outcome: Change From Baseline in H2O Detrusor Pressure at First Contraction at 6 Weeks
Description: Detrusor pressure was measured by means of urodynamic assessment (cystometry) for up to 6 weeks. Missing data were imputed by last observation carried forward (LOCF).
Time Frame: baseline and up to 6 weeks of treatment LOCF
Population: Modified intent-to-treat (mITT) population: participants included in the safety sample (received at least one dose), randomized correctly according to the Urodynamic Adjudication Board (UDAB), having one valid baseline and one valid (UDAB) on treatment urodynamic measurement. The number is not identical to participants who "completed" the study.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 119 | 135
millimeters of mercury (mmHg) | 0.085 (2.5821) | 0.743 (2.4199)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; ANCOVA models used for the secondary efficacy variables were the models determined for the primary efficacy variable or co-primary efficacy variable depending on the type of variable; Test type: Superiority or Other; p = 0.8533, ANCOVA — P-values were reported as nominal values and without any adjustments for multiplicity; Mean Difference (Final Values) = 0.657, 95% CI [-6.335 to 7.650] — Placebo- Vardenafil

4. Secondary Outcome: Change From Baseline in Volume at First Detectable Leakage at 6 Weeks
Description: First detectable leakage was determined by means of cystometry as an obligatory urodynamic measure. Missing data was imputed by last observation carried forward (LOCF).
Time Frame: baseline and up to 6 weeks of treatment LOCF
Population: Modified intent-to-treat (mITT): participants included in the safety sample (received at least one dose), randomized correctly according to the Urodynamic Adjudication Board (UDAB), having one valid baseline and one valid (UDAB) on treatment urodynamic measurement. The number is not identical to participants who "completed" the study.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 121 | 134
mL | 42.307 (7.9013) | 26.717 (7.5039)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1539, ANCOVA — P-values were reported as nominal values and without any adjustments for multiplicity; Mean Difference (Final Values) = -15.590, 95% CI [-37.057 to 5.876] — Placebo- Vardenafil

5. Secondary Outcome: Change From Baseline in Maximum Cystometric Bladder Capacity at 6 Weeks
Description: Maximum cystometric bladder capacity was defined as the volume at which either significant leakage or discomfort/pain occurred. Missing data were imputed by last observation carried forward (LOCF).
Time Frame: baseline and up to 6 weeks of treatment LOCF
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 125 | 136
mL | 40.274 (7.4986) | 27.900 (7.1839)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2348, ANCOVA — P-values were reported as nominal values and without any adjustments for multiplicity; Mean Difference (Final Values) = -12.374, 95% CI [-32.834 to 8.087] — placebo - vardenafil

6. Secondary Outcome: Change From Baseline in Volume at First Desire to Void at 6 Weeks
Description: Volume at first desire to void was recorded during urodynamic assessments. Missing data were imputed by last observation carried forward (LOCF).
Time Frame: baseline and up to 6 weeks of treatment LOCF
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 125 | 136
mL | 30.655 (6.0503) | 22.460 (5.7959)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3289, ANCOVA — P-values were reported as nominal values and without any adjustments for multiplicity; Mean Difference (Final Values) = -8.195, 95% CI [-24.692 to 8.303] — placebo - vardenafil

7. Secondary Outcome: Change From Baseline in Average Number of Urgencies Per Day at 6 Weeks
Description: The average number of urgencies was derived from the number of urgencies reported by the participants in a 7 day micturition diary. Missing data were imputed by last observation carried forward.
Time Frame: baseline and up to 6 weeks of treatment LOCF
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: urgencies per day
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 163 | 178
urgencies per day | -1.861 (0.2768) | -1.139 (0.2658)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0609, ANCOVA — P-values were reported as nominal values and without any adjustments for multiplicity; Mean Difference (Final Values) = 0.721, 95% CI [-0.033 to 1.476] — placebo - vardenafil

8. Secondary Outcome: Change From Baseline in Average Number of Daily Involuntary Discharges of Urine at 6 Weeks
Description: The average number of daily involuntary discharges of urine was derived from the number of discharges reported by the participants in a 7 day micturition diary. Missing data were imputed by last observation carried forward.
Time Frame: baseline and up to 6 weeks of treatment LOCF
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: involuntary discharges per day
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 162 | 178
involuntary discharges per day | -0.566 (0.1241) | 0.447 (0.1188)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4928, ANCOVA — P-values were reported as nominal values and without any adjustments for multiplicity; Mean Difference (Final Values) = 0.118, 95% CI [-0.220 to 0.456] — placebo - vardenafil

9. Secondary Outcome: Change From Baseline in Peak Urinary Flow at 6 Weeks in Men Aged 50 Years and Older
Description: Peak urinary flow (Qmax) was measured using urodynamic assessments (voiding / flow cystometry) for up to 6 weeks. Missing data were imputed by last observation carried forward (LOCF).
Time Frame: baseline and up to 6 weeks of treatment LOCF
Population: mITT: Participants who received at least one dose, randomized correctly according to Urodynamic Adjudication Board (UDAB), having one valid baseline and one valid (UDAB) on treatment urodynamic measurement. Qmax is based on men predominantly aged 50 years and older but includes a few males who had Qmax collected even if younger than 50 years.
Measure: Least Squares Mean (Standard Error); unit: milliliter per second (mL/s)
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 39 | 55
milliliter per second (mL/s) | 1.129 (0.6301) | 0.306 (0.5351)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3248, ANCOVA — P-values were reported as nominal values and without any adjustments for multiplicity; Mean Difference (Final Values) = -0.823, 95% CI [-2.476 to 0.829] — placebo - vardenafil

10. Secondary Outcome: Change From Baseline in the Total Score of the Overactive Bladder Questionnaire (OAB-q) at 6 Weeks
Description: The OAB-q is a validated, self-administered questionnaire that quantifies bladder symptoms and quality of life. It comprises 33 items (6-point scale for each item). The total score ranges from 33 (minimum symptoms) to 198 (maximum symptoms). On each item, participants provide their rating over the past 4 weeks. Missing data were imputed by LOCF.
Time Frame: baseline and up to 6 weeks of treatment LOCF
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Number analyzed (Participants) | 156 | 169
scores on a scale | 8.929 (1.2627) | 7.834 (1.2181)
Statistical Analysis 1: Comparison: Vardenafil HCl (Levitra, BAY38-9456) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.5312, ANCOVA — P-values were reported as nominal values and without any adjustments for multiplicity; Mean Difference (Final Values) = -1.095, 95% CI [-4.533 to 2.342]

ADVERSE EVENTS:
Arm/Group | Vardenafil HCl (Levitra, BAY38-9456) | Placebo
Serious Adverse Events (participants affected / at risk) | 4/198 | 4/198
Other Adverse Events (participants affected / at risk) | 78/198 | 39/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vardenafil HCl (Levitra, BAY38-9456) (N=198) | Placebo (N=198)
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vardenafil HCl (Levitra, BAY38-9456) (N=198) | Placebo (N=198)
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Dyspepsia (Gastrointestinal disorders) | 10 | 1
Flatulence (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 5 | 4
Asthenia (General disorders) | 4 | 0
Fatigue (General disorders) | 7 | 3
Urinary tract infection (Infections and infestations) | 8 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 1
Dizziness (Nervous system disorders) | 8 | 4
Headache (Nervous system disorders) | 37 | 18
Flushing (Vascular disorders) | 5 | 1
Hot flush (Vascular disorders) | 2 | 4

LIMITATIONS AND CAVEATS:
635 participants were screened; 238 were not randomized because they did not fulfill the inclusion/exclusion criteria. Cystometric bladder compliance not presented since only relevant to characterization of detrusor overactivity, not to efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publishing incl confidential information only after Bayer written approval. Manuscript to Bayer 60 days before submission. Confidential Information to be deleted. Other Bayer comments to be considered, if they do not alter the scientific character. If no Bayer comment within 45 days, consider approval given. If multisite study Principal Investigator (PI) not to independently publish results before publication of multisite paper, but PI not restricted from 24 months from study completion onwards.